CLINICAL TRIAL: NCT04047459
Title: Identification of Novel Genes Involved in Cancer Cell Extravasation by Transcriptional Profiling of Primary Organ-specific Endothelial Cells and in Vitro 3D Models
Brief Title: Investigation of Cancer Cell Extravasation Through mRNA Analysis of Organ-specific Endothelial Cells and Microfluidics
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: BRCP USA
Record Dates: First submitted 2017-12-06; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer Metastatic
Keywords: Organ specific endothelium; Microfluidics; Cancer cell extravasation
MeSH Terms: interventions — Cell Separation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of bone and muscle tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient undergoing prosthetic surgery: Patients undergoing surgery for the insertion of a hip prosthesis or a cruciate ligament reconstruction will be included. On those patients tissue samples collection and cells isolation will be performed
  Interventions: Other: Tissue samples collection and cells isolation

INTERVENTIONS:
Other: Tissue samples collection and cells isolation — During surgery, leftover samples of bone (femoral head/ trabecular bone tissue) and muscle will be collected. Then they will be sent to the laboratory where isolation of cells will be performed.

SUMMARY:
The project aims at unraveling the role of organ-specific endothelia mediating the preferential metastasisation of breast cancer cells to bone by using a multi-faceted approach, integrating microfluidics and transcriptomic profiling. Based on a recently study published by the investigators [Jeon et al., PNAS 2015], it can be hypothesized that phenotypic differences at the level of organ-specific endothelial cells are able to drive the preferential extravasation of breast cancer cells to specific sites. Hence, the transcriptional profile of primary organ-specific endothelial cells derived from healthy patients (i.e. non-affected by breast cancer) will be analyzed to identify phenotypic differences between organ-specific populations of endothelial cells. These analyses will allow to identify potential target genes involved in the organ-specific extravasation of cancer cells (i.e. genes differentially expressed by endothelia of preferential and non-preferential metastasisation sites). The selected genes will be silenced and the effect of gene silencing will be evaluated through microfluidic in vitro organ-specific 3D models designed to study cancer cell extravasation.

DETAILED DESCRIPTION:
In particular, the main aim of the study will be to highlight differences between bone and skeletal muscle microenvironments, which are respectively preferential and non-preferential metastasisation sites for breast cancer cells, in order to identify specific pathways driving breast cancer cells extravasation. To this purpose, differences in the transcriptional profile of ECs derived from bone and muscle endothelium will be investigated. These analyses will be used to select target genes differentially expressed by bone- and muscle-specific ECs. Then, ECs obtained from bone and muscle endothelium will be respectively used to mimic bone and muscle microvessel environments in microfluidic in vitro 3D models allowing for the study of breast cancer cell extravasation. The genes selected according to the results of the transcriptomic analysis (e.g. genes expressed in ECs derived from bone endothelium, but not expressed in ECs derived from muscle endothelium) will be silenced and the effect of gene silencing will be evaluated monitoring breast cancer cell extravasation in order to verify the involvement of the selected genes in this process.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65 years
* patients undergoing cruciate ligament surgery or hip arthroplasty
* subscription of informed consent

Exclusion Criteria:

- HIV, HCV, HBV, TPHA viral

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing hip or knee surgery, from whom samples of waste bone and muscle tissues can be harvested.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Genes differentially expressed by bone and muscle ECs | 31/05/2018
  Differential expression of genes will be determined by transcriptomic analysis of mRNA (with genome-wide mRNA array tools) derived from bone and muscle ECs

SECONDARY OUTCOMES:
Differences in adhesive properties of bone and muscle ECs | 31/05/2018
  Bone and muscle derived ECs will be compared in terms of immunofluorescent staining for adhesion molecules (ICAM-1, E-selectin)
Differences in cell adhesion between bone and muscle ECs | 31/05/2018
  Bone and muscle derived ECs will be compared in terms of number of cells adhered (neutrophils, ...)
Differences in angiogenic potential between bone and muscle ECs | 31/05/2018
  Bone and muscle derived ECs will be compared in terms of angiogenic sprouting, by analyzing immunofluorescence images
Selection of potential target genes involved in breast cancer metastasis | 31/05/2018
  Differentially expressed genes potentially involved in breast cancer cells extravasation and metastasis formation

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Moretti, PhD, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Galeazzi Orthopedic Hospital, Milan, Italy